CLINICAL TRIAL: NCT03068689
Title: Remote Ischaemic PreConditioning (RIPC) in Partial Nephrectomy for the Prevention of Ischemia/Reperfusion Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RIPC
Record Dates: First submitted 2017-02-22; First posted 2017-03-03 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Reperfusion Injury
Keywords: Partial nephrectomy, RIPC, Reperfusion Injury
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (RIPC) (Experimental): RIPC treatment prior to partial nephrectomy.
  Interventions: Procedure: RIPC
- Placebo Control (Placebo Comparator): Placebo prior to partial nephrectomy.
  Interventions: Other: Placebo

INTERVENTIONS:
Procedure: RIPC — RIPC is delivered with a standard blood pressure cuff placed on the upper arm and another standard blood pressure cuff placed on the upper thigh. The cuffs are then simultaneously inflated to 200 mm HG and left inflated for 5 minutes, then deflated to 0 mmHG and left uninflated for 5 minutes. This cycle is repeated twice, so that the RIPC protocol takes 20 minutes in total. If the systolic blood pressure is > 185mm HG the cuffs are inflated to 15 mmHG above that level.
  Arms: Intervention (RIPC)
Other: Placebo — Placebo
  Arms: Placebo Control

SUMMARY:
"Remote Ischaemic PreConditioning" (RIPC) is performed prior to partial nephrectomy. Postoperative calprotectin dynamics and Blood Oxygen-Level-Dependent (BOLD) MRI are used to to demonstrate the potential renoprotective effect of RIPC

DETAILED DESCRIPTION:
Partial nephrectomy represents the gold standard in organ sparing kidney surgery. Cold ischaemia prevents major bleeding but can yet be associated with impaired kidney function due to reperfusion injury to the tubuli.

Patients undergoing partial nephrectomy (any surgical technique, open, retroperitoneoscopic, transperitoneal, Da Vinci assisted) will be treated with "Remote Ischaemic PreConditioning" (RIPC). RIPC is delivered with a standard blood pressure cuff placed on the upper arm and another standard blood pressure cuff placed on the upper thigh. The cuffs are then simultaneously inflated to 200 mm HG and left inflated for 5 minutes, then deflated to 0 mmHG and left uninflated for 5 minutes. This cycle is repeated twice, so that the RIPC protocol takes 20 minutes in total. If the systolic blood pressure is > 185mm HG the cuffs are inflated to 15 mmHG above that level. Several studies already demonstrated the reno- and cardioprotective potential of "Remote Ischaemic PreConditioning" (RIPC). It was shown that urinary calprotectin can be used to monitor tubular damage after nephron sparing surgery. Postoperative calprotectin dynamics will be monitored in order to demonstrate the potential renoprotective effect of RIPC. Additionally a BOLD MRI will be performed to to visualize ischemia/reperfusion injury.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Kidney tumor (any entity, benign, malign)
* Partial nephrectomy (any surgical technique, open, retroperitoneoscopic, transperitoneal, Da Vinci assisted)
* 18 years of age
* Sufficient perfusion of all 4 extremities
* palpable distal pulses: A. radialis and A. dorsalis pedis or A.tibialis post.

Exclusion Criteria:

* Women who are pregnant
* Significant peripheral arterial disease affecting upper and/or lower limbs or history of
* Significant renal disease (GFR <15 ml/min/1.73m2) or undergoing haemodialysis
* Concomitant therapy with glibenclamide or nicorandil (due to potential inference with RIPC)
* Urothelial cancer
* Acute Urinary tract infection
* international normalized ratio (INR) >2 (haematoma risk at cuff site)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Biomarker reduction | Baseline, 5 days and 3 months
  The study seeks primarily to determine the reduction of the biomarker concentration (Calprotectin and NGAL) in urine. Change in biomarkers will be measured at baseline, during 5 days after surgery and at timepoint month 3.

SECONDARY OUTCOMES:
Acute renal failure | Baseline, 5 days, 3 Months
  The secondary objective is to demonstrate the effect/reduction acute renal failure after RIPC as compared to the control group.
  Number of patients with acute renal failure will be compared between both groups.
  Acute renal failure will be assessed in the days after surgery (acute kidney failure)
Chronic renal failure | Baseline, 3 Months
  Number of patients with chronic renal failure will be compared between both groups.
  Chronic renal failure will be assessed in at baseline until timepoint month 3 (chronic kidney failure).
Tubular damage in BOLD MRT | Baseline, day 2
  Δ R2*-values in BOLD magnetic resonance tomography (MRT) will be compared between both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Ebbing, MD, Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Clinic of Urology, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No